CLINICAL TRIAL: NCT00044252
Title: Role of Serum Gonadal and Neuroactive Steroids in the Seizure Susceptibility of Women With Catamenial Epilepsy
Brief Title: Role of Hormones in Susceptibility to Seizures in Women With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020256; 02-N-0256
Record Dates: First submitted 2002-08-22; First posted 2002-08-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-01-22

CONDITIONS: Epilepsy
Keywords: Neurosteroids; Complex Partial Seizure; Menstrual Cycle; Allopregnanolone; Catamenial Epilepsy; Seizures; Epilepsy; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Epilepsy; Seizures

SUMMARY:
This study will measure and compare hormone levels in women with catamenial epilepsy (epilepsy in which seizures are more frequent during menstrual periods), women with seizures not related to their menstrual cycle, and normal control subjects. It will determine whether there are differences among the three groups in their hormone levels or in how fast the levels change. It will also examine what relationship, if any, exists between hormone changes and seizures in women with catamenial epilepsy. The hormones under study include the gonadal hormones estrone, estradiol and progesterone, and the neuroactive steroids allopregnanolone, pregnenolone, and dehydroepiandrosterone.

Women who meet the following criteria may be eligible for this 3-month study:

* Between 18 and 45 years of age, with catamenial epilepsy
* Between 18 and 45 years of age, with seizures, but not catamenial epilepsy
* Between 18 and 45 years of age, without seizures

All participants will have a physical examination at the beginning of the study, at each clinic visit, and at completion or withdrawal from the study. In addition, they will undergo the following procedures:

Baseline Monitoring

For the first 2 months, all participants will keep a diary of their temperature and onset of menses. Women with epilepsy will also record their seizures.

Electroencephalography (EEG)

Healthy volunteers will have a 45-minute EEG (recording of the electrical activity of the brain) at the beginning of each menstrual cycle and each day during the menses. Women with epilepsy will have continuous EEG monitoring for 8 days, beginning 5 days before their menstrual period is expected. The continuous monitoring can be done on an outpatient basis, using a portable EEG recording device, or as an inpatient, with admission to the hospital for the 8 days of recording.

Blood Sampling

All participants will have a small blood sample (2 teaspoons) drawn once a day on days 10, 14, 17, 19 and 21 of their menstrual cycle and three times a day on day 6 and for a period of 8 days, starting 5 days before the expected menses and continuing for 3 days of the next cycle. For the days with three blood draws, a small needle that can stay in place for up to 72 hours will be placed in the arm to avoid the discomfort of multiple needle sticks.

DETAILED DESCRIPTION:
Objectives. This is an initial pilot study to acquire information upon which a more specific, statistically rigorous follow-on investigation will be based. The objectives of the overall project are: (1) to compare the absolute levels and rates of change in levels of gonadal and neuroactive steroids in women with complex partial seizures and catamenial epilepsy with those of women with non-catamenial epilepsy and women volunteers without epilepsy, and (2) to determine if fluctuations in the levels of gonadal hormones (estrone, estradiol, progesterone) and neuroactive steroids (allopregnanolone, pregnenolone and dehydroepiandrosterone) correlate with seizure occurrence and the frequency of interictal spikes/wave discharges in women with catamenial seizure exacerbations.

Study Populations. Group A: adult women with complex partial seizures and catamenial exacerbations. Group B: adult women with complex partial seizures without catamenial seizure exacerbations. Group C: adult female volunteers without epilepsy.

Design. Subjects will undergo baseline monitoring of seizures and menses for two months prior to entry. Upon enrollment into the study, blood (10 ml) will be drawn for determinations of estradiol, estrone, progesterone, allopregnanolone, dehydroepiandrosterone (DHEA) and pregnenolone in all study populations once daily at 08:30 hr on menstrual cycle days, 10, 14, 17, 19 and 21; and three times daily at 08:30, 13:30 and 18:00 starting 5 days before expected menses and continuing for a total of 8 days as well as on menstrual cycle day 6. During 8 days starting 5 days before expected menses interictal spike activity and seizures will also be monitored continuously with EEG. Comparisons of the rates of change of hormone levels and spike and seizure frequency will be made using the time derivatives of fluctuations in hormone levels or hormone level ratios. Comparisons of time series data will be made using nonlinear regression with an arbitrary (cubic spine) model.

Outcome Parameters. The goal of this preliminary study is to obtain data regarding the fluctuation, during one menstrual cycle, of several hormones in epileptic and non-epileptic women of reproductive age. If the data show a relationship between (i) falling levels of plasma progesterone and allopregnanolone, (ii) increased levels of DHEA or pregnenolone or (iii) increased ratios of estrogen/progesterone, DHEA/progesterone, DHEA/allopregnanolone, pregnenolone/allopregnanolone and seizure manifestations and EEG documented interictal spike and seizure activity it would support the hypothesis that alterations in the levels of these steroid hormones are related to seizure exacerbations in women with catamenial epilepsy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group A subjects will be 8 women between 18 and 45 years of age who have complex partial seizures with Type 1 catamenial seizure exacerbation as previously defined.

Group B subjects will be 8 women between 18 and 45 years of age with complex partial seizures who do not meet the criteria for catamenial seizure exacerbations. The presence or absence of Type 1 catamenial seizure exacerbation will be documented by a standard seizure calendar self-reported for at least two consecutive menstrual cycles.

Patients receiving antiepileptic drug therapy will continue on their medications.

All subjects must agree to use double barrier contraceptives, have an intrauterine device in place or practice abstinence during the course of the study.

Patients will be recruited from the epilepsy patient population at the National Institutes of Health.

Subjects in groups A and B will be matched for seizure frequency. Volunteers will be matched with the subjects in group A by age. In this pilot study, no attempt will be made to match patients according to anticonvulsant medications.

The patient will be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study.

EXCLUSION CRITERIA:

Any of the following conditions are cause for exclusion from the study:

Any illness requiring chronic drug therapy other than antiepileptic drugs.

Any history of an illness likely to be adversely affected by the trial.

Psychiatric hospitalization lasting more than 2 months at any time prior to the study.

Use of tricyclic antidepressants within 4 weeks prior to randomization and/or anti-psychotic drugs within 2 weeks prior to randomization.

Children will not be included in this pilot study, because the profile of hormonal secretion undergoes profound changes during puberty.

Use of illicit drugs, alcoholism or binge drinking as per medical history inventory.

Women who are unwilling to use an alternative to oral contraceptives for contraception, (double barrier contraceptives, intrauterine device or abstinence), and establish that they are currently not pregnant by submitting to a pregnancy test.

Exposure to any other investigational drug within 12 weeks prior to randomization.

Any history of endocrine dysfunction.

Women will be excluded if they do not have regular menstrual cycle intervals between 27 and 32 days or if they are pregnant, nursing or taking oral contraceptives or other reproductive hormones.

If a need should arise to change the antiepileptic regime during the study this subject will be excluded and replaced with another patient.

Women currently taking Phenobarbital or another barbiturate.

Women who are unwilling to refrain from strenuous exercise during the study.

Women who are unwilling to refrain from usage of herbal and soy products.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2002-07-26; Study Completion 2008-01-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Herzog AG, Klein P, Ransil BJ. Three patterns of catamenial epilepsy. Epilepsia. 1997 Oct;38(10):1082-8. doi: 10.1111/j.1528-1157.1997.tb01197.x. PMID 9579954